CLINICAL TRIAL: NCT05580744
Title: Effects of Augmented-reality Based Mirror Therapy on Sensorimotor Function of Upper Extremity
Brief Title: Augmented-reality Based Mirror Therapy in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-ER-111-246
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Rehabilitation; Technology; Mirror Movement Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Traditional occupational therapy (Active Comparator): Traditional occupational therapy delivered skill training related to daily living tasks.
  Interventions: Other: Traditional occupational therapy
- Mirror therapy using a mirror box (Active Comparator): Exercise of mirror therapy included movements of forearm, wrist, fingers and thumb, as well as a tendon gliding exercise using a mirror box .
  Interventions: Other: Mirror therapy using a mirror box
- Augmented reality-based mirror therapy (Experimental): Exercise of augmented reality-based mirror therapy included movements of forearm, wrist, fingers and thumb, as well as a tendon gliding exercise using an augmented reality mirror therapy system
  .
  Interventions: Other: Augmented reality-based mirror therapy

INTERVENTIONS:
Other: Traditional occupational therapy — Motor training targeted to goals that are relevant to the functional needs of the patient
  Arms: Traditional occupational therapy
Other: Mirror therapy using a mirror box — Mirror therapy using a mirror box
  Arms: Mirror therapy using a mirror box
Other: Augmented reality-based mirror therapy — Augmented reality-based mirror therapy
  Arms: Augmented reality-based mirror therapy

SUMMARY:
In the proposed study, the investigators assumed that mirror therapy combined with augmented reality technology will provide a better treatment effects than traditional mirror therapy for the patients with unilateral stroke. The aim of the study is to examine the difference in the treatment effects among the combination of task-oriented training with either augmented reality based mirror therapy, mirror therapy or traditional occupational therapy on the upper extremity function and brain activity of the stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke with unilateral side involved;
* A score of Mini-mental state examination greater than 24 for proving higher mental function
* Time of onset > 6 months before treatment begins; and
* Premorbid right-handedness.

Exclusion Criteria:

* Severe vision impairment;
* Major cognitive-perceptual deficit;
* Other brain disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Change in the result of Fugl-Meyer assessment (FMA) for motor function of upper extremity test | baseline, 9 weeks and 21 weeks
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.

SECONDARY OUTCOMES:
Change in the result of Modified Ashworth scale (MAS) | baseline, 9 weeks and 21 weeks
  Muscle tone is defined by the resistance of a muscle being stretched without resistance. The MAS scores were distributed across the entire scale, ranging from 0 to 4, that is convenient for the clinician use. The grading of the scale is described as below: 0) no increase in muscle tone; 1) minimal resistance at the end of the range of motion; 1+) slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the reminder (less than half) of the ROM; 2) more marked increase in tone but only after part is easily flexed; 3) considerable increase in tone; and 4) passive movement is difficult and affected part is rigid in flexion or extension.
Change in the result of Box and blocks test | baseline, 9 weeks and 21 weeks
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, 9 weeks and 21 weeks
  The Semmes-Weinstein monofilamenttest examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome.
Change in the result of Motor Activity Log | baseline, 9 weeks and 21 weeks
  Semi-structured interview examine how much and how well the subject uses their more-affected arm for 30 ADLs. Score range from 0-5. Higher values represent a better outcome.

OTHER OUTCOMES:
changes in oxygenated (HbO) and deoxygenated (Hb) hemoglobin concentrations using near infrared spectroscopy (NIRS) | baseline, 9 weeks and 21 weeks
  To investigate the activation of specific brain regions

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No